CLINICAL TRIAL: NCT04224480
Title: Longitudinal Immune-phenotyping of Surgically Resected HCC Following Neoadjuvant and Adjuvant Treatment With MK-3475
Brief Title: Longitudinal Immune-phenotyping of HCC Following MK-3475
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCS-OTSP-HCC1
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Neoadjuvant treatment will consist of one dose of IV pembrolizumab. Tumor resection will be performed approximately 4 weeks after neoadjuvant pembrolizumab. Adjuvant treatment with pembrolizumab will be administered 4 weeks after the surgery.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg of intravenous infusion every 3 weeks
  Other Names: MK-3475

SUMMARY:
The study comprises a main study of pembro-treated HCC patients and a sub-study of untreated HCC patients. In the main study, patients will be treated with pembrolizumab as neoadjuvant treatment approximately 4 weeks prior scheduled surgery. Adjuvant treatment with pembrolizumab with commence at approximately 4 weeks post-surgery for up to 12 months. Subjects will be followed up for a further 12 months after end of treatment for recurrence and survival.

The sub-study is a tumour sample collection study which will provide pre-treatment immune microenvironment data from up to 15 pairs of HCC/adjuvant liver tissue samples. Translational analyses performed for liver tissue samples in the sub-study will be harmonized with the analyses on liver tissue samples collected in the main study.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial. The subject may also provide consent for donation of tissue to the SingHealth Tissue Repository (STR). However, the subject may participate in the trial without participating in STR.
* Be male or female subject, who is at least 21 years of age on the date of first signed written informed consent
* Have diagnosis of HCC by AASLD imaging criteria or by cytology/histology.
* Have technically resectable HCC, with complete extirpation of HCC at end of surgery by resection +/- intra-operative radiofrequency ablation (RFA) at time of enrolment:

  * Without extrahepatic metastases

    * Regional lymph nodes (LN) <2 cm
    * Lung lesions <1 cm
  * Without invasion of main portal vein (PV3), or major left and right branches (PV2)
  * Future liver remnant of >40%
  * <5 hepatic lesions in total
* Have tumor larger than 1.5 cm in size
* Demonstrate adequate organ function as defined in Table 3, all screening labs should be performed within 14 days of neoadjuvant treatment initiation.

  * Absolute neutrophil count (ANC): ≥1,200/mcL
  * Platelets: ≥80,000/ mcL
  * Hemoglobin: ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
  * Serum creatinine: ≤1.5 X upper limit of normal (ULN) OR creatinine ≥60mL/min for subjects with creatinine >1.5X institutional ULN
  * Serum total bilirubin: ≤ 1.5 X ULN
  * AST (SGOT) and ALT (SGPT): ≤5.0 X ULN
  * Albumin: ≥3.0 g/dL
  * International Normalized Ratio (INR) or Prothrombin Time (PT) AND Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN OR within therapeutic range for subjects on anticoagulant therapy. Abnormalities will be corrected prior to liver resection, if necessary according to institution practice
* Have Child-Pugh score ≤ 6.
* Be scheduled for liver resection within 5-6 weeks.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Have a performance status of 0-1 using the ECOG Performance Scale.
* Have not had treatment for HCV or are not on current anti-HCV treatment for subjects with chronic infection by HCV. For subjects who have had anti-HCV therapy, the last dose of anti-HCV medication should be at least 4 weeks before first dose of pembrolizumab.
* Have HBV viral load under 100 IU/mL with or without treatment, for subjects with chronic hepatitis B infection. HBV viral load must be less than 100 IU/mL on at least 4 weeks of anti-viral therapy prior to first dose of pembrolizumab. Subjects on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study treatment. Subjects who are anti-HBc (+), negative for HBs Ag, negative for anti-HBs, and have an HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Protocol Chairperson. Physiologic dose of corticosteroid is defined as ≤ 10 mg/day prednisolone or equivalent.
* Has macrovascular invasion and distant metastases. Definition of metastases includes lymph nodes (LN) ≥ 2 cm in widest diameter and lung lesions ≥ 1 cm in widest diameter).
* Has tumor thrombus involvement in main portal vein (PV3), or major left and right branches (PV2) on pre-operative imaging.
* Has a recurrent HCC < 24 months after previous resection.
* Has had major surgery to any site within 4 weeks prior to the first dose of study drug.
* Has future liver remnant ≤ 40%.
* Has more than 5 lesions in total.
* Has encephalopathy.
* Has history of allergic disease or reactions likely to be exacerbated by any component of pembrolizumab.
* Has had a solid organ or hematologic transplant.
* Has had untreated esophageal or gastric variceal bleeding within the last 6 months.
* Has clinically apparent ascites on physical examination.
* Has had prior anti-cancer treatment for HCC, except for complete ablation of HCC by liver resection and/or RFA at least 24 months prior to current HCC diagnosis. Anti-cancer treatment includes but is not limited to loco-regional therapy (e.g. TACE, radiotherapy, immunotherapy, chemotherapy or neoadjuvant therapy).
* Has previous or concomitant malignancies at other sites, except effectively treated non-melanoma carcinoma of the skin or in situ cervical cancer or effectively treated malignancy that has been in remission for more than 5 years and is highly likely to have been cured.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or any uncontrolled arrhythmia at the time of enrollment into study.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including dialysis.
* Has known psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with trial procedures.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or if the subject has previously participated in Merck pembrolizumab clinical trials
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Is currently participating, or has participated, in a study of an investigational agent and received study therapy, herbal/complementary oral or IV medicine, or used an investigation device within 4 weeks of the first dose of treatment. Subjects must also have recovered from associated therapy (i.e. to Grade ≤ 1 or baseline) and from AEs due to any prior therapy.
* Has had a minor surgery ≤ 7 days prior to the first dose of study treatment (Cycle 1, Day 1).
* Has an active infection requiring systemic therapy.
* Has dual active HBV infection [HBsAg (+) and/or detectable HBV DNA] and HCV infection [anti-HCV Ab (+) and detectable HCV RNA] at study entry.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with HCC recurrence | 2 years after hepatic resection
  To evaluate the effect of neoadjuvant and adjuvant pembrolizumab on recurrence rate
Number of CD8+ Ki67+ T cells found in resected tumour from subjects | Up to 24 months after hepatic resection
  To compare the phenotype of immune cells in the tumor microenvironment after tumor resection from recurrence-free verses recurrent subjects receiving pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Han Chong Toh, MD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gao Q, Wang XY, Qiu SJ, Yamato I, Sho M, Nakajima Y, Zhou J, Li BZ, Shi YH, Xiao YS, Xu Y, Fan J. Overexpression of PD-L1 significantly associates with tumor aggressiveness and postoperative recurrence in human hepatocellular carcinoma. Clin Cancer Res. 2009 Feb 1;15(3):971-9. doi: 10.1158/1078-0432.CCR-08-1608. PMID 19188168
- [Background] Welker MW, Bechstein WO, Zeuzem S, Trojan J. Recurrent hepatocellular carcinoma after liver transplantation - an emerging clinical challenge. Transpl Int. 2013 Feb;26(2):109-18. doi: 10.1111/j.1432-2277.2012.01562.x. Epub 2012 Sep 21. PMID 22994652